CLINICAL TRIAL: NCT02848963
Title: Effect of Ketamine-propofol Mixture on Postoperative Pain and Sedation-agitation
Brief Title: Comparison of Ketamine-propofol Combinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Ketamine-Propofol
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-10

CONDITIONS: Agitation; Postoperative Pain
MeSH Terms: conditions — Psychomotor Agitation; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ketamine-propofol mixture 5/1 (Active Comparator): Ketamine-propofol mixture will be compare for every groups.
  Interventions: Drug: Ketamine-propofol mixture
- ketamine-propofol mixture 10/1 (Active Comparator): Ketamine-propofol mixture will be compare for every groups.
  Interventions: Drug: Ketamine-propofol mixture
- Ketamine-propofol mixture 6,7/1 (Active Comparator): Ketamine-propofol mixture will be compare for every groups
  Interventions: Drug: Ketamine-propofol mixture

INTERVENTIONS:
Drug: Ketamine-propofol mixture — Ratio of Ketamine-propofol mixture will be compare for every groups.
  Other Names: ketofol

SUMMARY:
ASA I-II 3-12 years old children participated to this study. All Participants will divide into the three groups. In Groups I, 2,5 mg/kg propofol and 0,5 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 5/1 ratio of ketamine-propofol mixture with %67 of Mcfarlan dose regiment.

In Groups II, 2,75 mg/kg propofol and 0,41 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 6,7/1 ratio of ketamine-propofol mixture with %80 of Mcfarlan dose regiment.

In Groups III, 3 mg/kg propofol and 0,3 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 10/1 ratio of ketamine-propofol mixture with %90 of Mcfarlan dose regiment.

After than surgical operation recovery time, PAED scores, FLACC scores, Staying time in PACU will be recorded. These data will be evaluated with statistically.

DETAILED DESCRIPTION:
ASA I-II, 3-12 years old children who will operate due to tonsillectomy and adenoidectomy. will be participated in to this study. All Participants will divide into the three groups. In Groups I, 2,5 mg/kg propofol and 0,5 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 5/1 ratio of ketamine-propofol mixture with %67 of Mcfarlan dose regiment.

In Groups II, 2,75 mg/kg propofol and 0,41 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 6,7/1 ratio of ketamine-propofol mixture with %80 of Mcfarlan dose regiment.

In Groups III, 3 mg/kg propofol and 0,3 mg/kg ketamine will apply at anaesthesia induction. General anaesthesia will be performed with 10/1 ratio of ketamine-propofol mixture with %90 of Mcfarlan dose regiment.

McFarlan dose regiments include 15 mg/kg/h infusion during 15 minutes, 13 mg/kg/h infusion during second 15 minutes, 11 mg/kg/h infusion from 30 to 60 minutes, 10 mg/kg/h from 1 to 2 h.

Anaesthesia dept will be detect with BIS monitoring during operation. After than surgical operation recovery time, PAED scores, FLACC scores, staying time in PACU and extubation time will be record. At the end of the study, these data will be evaluated with statistically.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II children
* Children who will be performed to adenoidectomy and tonsillectomy surgical operations

Exclusion Criteria:

* ASA III-IV children
* Patients over the age of 13

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PAED(Paediatric Anaesthesia Emergence Delirium) Scores Evaluation | During 1 hour at post operative period
  All patients will be evaluate with PAED scores at PACU during first 1 hour

SECONDARY OUTCOMES:
Anaesthesia depth assessed using the Bispectral Index (BIS) | During peroperative period.
  All Patients will monitored with BIS monitoring during operation.
Extubation time | time from injection of reversal to extubation, through patient extubated
  At the end of the surgery, time from injection of reversal to extubation
FLACC(Face, leg movement, activity, craying, consolability) | During 1 hour at post operative period
  All patients will be evaluate with FLACC scores at PACU during first 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Özcengiz, Professor, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biricik E, Karacaer F, Gulec E, Surmelioglu O, Ilginel M, Ozcengiz D. Comparison of TIVA with different combinations of ketamine-propofol mixtures in pediatric patients. J Anesth. 2018 Feb;32(1):104-111. doi: 10.1007/s00540-017-2438-8. Epub 2017 Dec 16. PMID 29249041